CLINICAL TRIAL: NCT05650294
Title: Investigation of Uptake of Two Different Omega-3 Fatty Acid Products in Healthy Subjects - a Randomized, Two-way Cross-over Study
Brief Title: Uptake of an Omega-3 Oil in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aker BioMarine Human Ingredients AS (Industry)
Collaborators: BioTeSys GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: BTS1879/22 // AKBM188H
Record Dates: First submitted 2022-11-24; First posted 2022-12-14 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-03

CONDITIONS: Absorption; Pharmacokinetics
Keywords: Omega 3 fatty acids; EPA; DHA

STUDY DESIGN:
Intervention Model Description: randomized, two-way cross-over study
Masking Description: The clinical study will be performed unblinded. However, analysis of blood samples at analysis partner will be performed blinded. After closure of data base, data will be unblinded and evaluated according to product affiliation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active group (Active Comparator): This group will receive a single dose of the PL+ omega 3 fatty acids capsules first, then receive a single dose of the standard FO EE omega 3 fatty acids capsules. Wash-out period is 2 weeks between treatments.
  Interventions: Dietary Supplement: PL+ omega 3 fatty acids; Dietary Supplement: FO EE fatty acids
- Placebo group (Placebo Comparator): This group will receive a single dose of the standard FO EE omega 3 fatty acids capsules first, then receive a single dose of the PL+ omega 3 fatty acids capsules. Wash-out period is 2 weeks between treatments.
  Interventions: Dietary Supplement: PL+ omega 3 fatty acids; Dietary Supplement: FO EE fatty acids

INTERVENTIONS:
Dietary Supplement: PL+ omega 3 fatty acids — PL+ omega 3 fatty acids is a food supplement that combines krill oil and FO EE. The dose will be around 1250 mg EPA+DHA.
Dietary Supplement: FO EE fatty acids — A conventional fish oil food supplement containing EPA and DHA in the EE form. The dose will be 1250 mg EPA+DHA.

SUMMARY:
The goal of this clinical trial is to compare the uptake of two different omega-3 fatty acid preparations in healthy adults. The main question it aims to answer is whether the two different preparations have the same uptake after single dose supplementation.

DETAILED DESCRIPTION:
Participants will be asked to take capsules of the new "phospholipids+" (PL+) omega-3 product (a combination product of krill oil and fish oil) in the morning with a low-fat breakfast. This product contains around 1250 mg eicosapentaenoic acid (EPA) + docosahexaenoic acid (DHA).

Researchers will compare this group with another group that takes standard fish oil (FO) ethyl esters (EE, with the same amount of EPA+DHA) to see if there are differences in pharmacokinetic parameters, including incremental area under the curve (iAUC), the maximum concentration of (Cmax) and the time it takes for EPA, DHA and EPA+DHA to reach the maximum concentration (Tmax) in plasma.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females (1:1) aged 18 - 65 years
* Capable and willing to give written informed consent, which includes compliance with the requirements and restrictions listed in the consent form
* Have a low habitual consumption of fatty fish and seafood, defined as a frequency of twice per month or less
* No fish consumption at least two weeks prior to screening visit
* Omega-3 index (≤ 7 %)
* Non-smoker
* BMI: 18 to 32 kg/m2

Exclusion Criteria:

* Omega-3 supplementation history within the last 4 weeks
* Have clinical evidence of significant unstable or uncontrolled acute or chronic diseases, i.e., diabetes, cardiovascular, pulmonary, hematologic, gastrointestinal, neurological, or infectious diseases which could confound the results of the study or put the subject at undue risk
* Have current drug or alcohol abuse or dependence, or a history of drug or alcohol abuse or dependence within 365 days prior to baseline
* Pregnancy, breast feeding or intention to become pregnant during the study (a pregnancy test will be conducted during screening and visits 1-2)
* General Safety & Laboratory Exclusion Criteria. Patients will be excluded from the study based on the following criteria:

  * Haemoglobin: < 12.0 g/dL (women); < 13.5 g/dL (men)
  * Platelets: < 150 x 103/μL
  * Leukocytes < 4,4 x 103/mm3
  * Aspartate transaminase (AST) or alanine transaminase (ALT) within the normal range
  * Serum creatine within the normal range
  * or further for this study clinically relevant abnormal laboratory findings at screening
* Significant changes in lifestyle or medication (within last 2 months)
* Chronic intake of substances affecting blood coagulation (e.g. acetylic acid, anticoagulants (e.g. Marcumar), diuretics, thiazides), which in the investigator's opinion would impact subject safety
* Difficulty swallowing capsules or predicted inability to swallow the study products
* Individuals who have made a blood donation in excess of 500 mL or who had excess blood loss within the 4 months before the study starts
* Individuals who are currently enrolled in an ongoing clinical trial or who have been an active participant in a clinical trial within the last 4 weeks
* A known allergy or hypersensitivity to any of the ingredients of the study products
* Not willing to abstain from fish consumption or foods/oils high in omega-3 fatty acids
* Subjects considered inappropriate for the study by investigators, including subjects who are unable or unwilling to show compliance with the protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2023-02-17 (Actual); Study Completion 2023-02-17 (Actual)

PRIMARY OUTCOMES:
Comparison of iAUC of EPA+DHA from 0 to 12 hours (iAUC0-12h) between two study products | 0h-12h (on Day 1 and Day 15)
  Blood concentrations of EPA + DHA in plasma at 0h and 12h will be analyzed, and determination of iAUC0-12h will be calculated. After getting the iAUC0-12h, difference of AUC curves between groups will be calculated.
  The time point 0h is defined as the time when study subjects is taking the supplement, while time point 12h is defined as 12 hours after the intake of supplement.

SECONDARY OUTCOMES:
Comparison of iAUC of EPA+DHA from 0 to 24hours (iAUC0-24h) between two study products | 0h-24h (on Day 2 and Day 16)
  Blood concentrations for EPA+DHA in plasma at 0h and 24h will be analyzed, and iAUC0-24h will be calculated. After getting the iAUC0-24h, difference of AUC curves between groups will be calculated.
  The time point 0h is defined as the time when study subjects is taking the supplement, while time point 24h is defined as 24 hours after the intake of supplement.
Comparison of iAUC EPA+DHA from 0 to 72hours (iAUC0-72h) between two study products | 0h-72h (on Day 4 and Day 18)
  Blood concentrations for EPA+DHA in plasma at 0h and 72h will be analyzed, and iAUC0-72h will be calculated. After getting the iAUC0-72h, difference of AUC curves between groups will be calculated.
  The time point 0h is defined as the time when study subjects is taking the supplement, while time point 72h is defined as 72 hours after the intake of supplement.
Comparison of iAUC EPA from 0 to 12hours (iAUC0-12h) between two study products | 0h-12h (on Day 1 and Day 15)
  Blood concentrations for EPA in plasma at 0h and 12h will be analyzed, and iAUC0-12h will be calculated. After getting the iAUC0-12h, difference of AUC curves between groups will be calculated.
  The time point 0h is defined as the time when study subjects is taking the supplement, while time point 12h is defined as 12 hours after the intake of supplement.
Comparison of iAUC DHA from 0 to 12hours (iAUC0-12h) between two study products | 0h-12h (on Day 1 and Day 15)
  Blood concentrations for DHA in plasma at 0h and 12h will be analyzed, and iAUC0-12h will be calculated. After getting the iAUC0-12h, difference of AUC curves between groups will be calculated.
  The time point 0h is defined as the time when study subjects is taking the supplement, while time point 12h is defined as 12 hours after the intake of supplement.
Comparison of iAUC EPA from 0 to 24hours (iAUC0-24h) between two study products | 0h-24h (on Day 2 and Day 16)
  Blood concentrations for EPA in plasma at 0h and 24h will be analyzed, and iAUC0-24h will be calculated. After getting the iAUC0-24h, difference of AUC curves between groups will be calculated.
  The time point 0h is defined as the time when study subjects is taking the supplement, while time point 24h is defined as 24 hours after the intake of supplement.
Comparison of iAUC DHA from 0 to 24hours (iAUC0-24h) between two study products | 0h-24h (on Day 2 and Day 16)
  Blood concentrations for DHA in plasma at 0h and 24h will be analyzed, and iAUC0-24h will be calculated. After getting the iAUC0-24h, difference of AUC curves between groups will be calculated.
  The time point 0h is defined as the time when study subjects is taking the supplement, while time point 24h is defined as 24 hours after the intake of supplement.
Comparison of iAUC EPA from 0 to 72hours (iAUC0-72h) between two study products | 0h-72h (on Day 4 and Day 18)
  Blood concentrations for EPA in plasma at 0h and 72h will be analyzed, and iAUC0-72h will be calculated. After getting the iAUC0-72h, difference of AUC curves between groups will be calculated.
  The time point 0h is defined as the time when study subjects is taking the supplement, while time point 72h is defined as 72 hours after the intake of supplement.
Comparison of iAUC DHA from 0 to 72hours (iAUC0-72h) between two study products | 0h-72h (on Day 4 and Day 18)
  Blood concentrations for DHA in plasma at 0h and 72h will be analyzed, and iAUC0-72h will be calculated. After getting the iAUC0-72h, difference of AUC curves between groups will be calculated.
  The time point 0h is defined as the time when study subjects is taking the supplement, while time point 72h is defined as 72 hours after the intake of supplement.
Difference on Cmax of EPA+DHA between two products | Day 1 and Day 15
  Cmax of EPA+DHA will be calculated for both products, and the difference will be compared between the products.
Difference on Cmax of EPA between two products | Day 1 and Day 15
  Cmax of EPA will be calculated for both products, and the difference will be compared between the products.
Difference on Cmax of DHA between two products | Day 1 and Day 15
  Cmax of DHA will be calculated for both products, and the difference will be compared between the products.
Difference on Tmax of EPA+DHA between two products | Day 1 and Day 15
  Tmax of EPA+DHA will be calculated for both products, and the difference will be compared between the products.
Difference on Tmax of EPA between two products | Day 1 and Day 15
  Tmax of EPA will be calculated for both products, and the difference will be compared between the products.
Difference on Tmax of DHA between two products | Day 1 and Day 15
  Tmax of DHA will be calculated for both products, and the difference will be compared between the products.
Difference on total omega 6 fatty acids vs total omega 3 fatty acid ratio (n-6/n-3) in plasma at 12 hours between two products | Day 1 and Day 15
  Total omega 6 fatty acids include: linoleic acid, γ-Linolenic acid, eicosadienoic acid, eicosatrienoic acid, arachidonic acid, adrenic acid, and docosapentaenoic acid. Total omega 3 fatty acids include: α-Linolenic acid, EPA, docosapentaenoate acid and DHA. The difference on n-6/n-3 ratio will be calculated between two products.
  The time point 12h is defined as 12 hours after the intake of supplement.
Difference on total omega 6 fatty acids vs total omega 3 fatty acid ratio (n-6/n-3) in plasma at 24 hours between two products | Day 2 and Day 16
  Total omega 6 fatty acids include: linoleic acid, γ-Linolenic acid, eicosadienoic acid, eicosatrienoic acid, arachidonic acid, adrenic acid, and docosapentaenoic acid. Total omega 3 fatty acids include: α-Linolenic acid, EPA, docosapentaenoate acid and DHA. The difference on n-6/n-3 ratio will be calculated between two products.
  The time point 24h is defined as 24 hours after the intake of supplement.
Difference on total omega 6 fatty acids vs total omega 3 fatty acid ratio (n-6/n-3) in plasma at 72 hours between two products | Day 4 and Day 18
  Total omega 6 fatty acids include: linoleic acid, γ-Linolenic acid, eicosadienoic acid, eicosatrienoic acid, arachidonic acid, adrenic acid, and docosapentaenoic acid. Total omega 3 fatty acids include: α-Linolenic acid, EPA, docosapentaenoate acid and DHA. The difference on n-6/n-3 ratio will be calculated between two products.
  The time point 72h is defined as 72 hours after the intake of supplement.

OTHER OUTCOMES:
Number of participants with treatment-related adverse events (AE) as assessed by Common Terminology Criteria for Adverse Events (CTCAE) v4.0 | Day 1 to Day 3 and Day 15 to Day 18
  During the study period, any changes in physical conditions will be evaluated by investigator using CTCAE v4.0 criteria and will be recorded as AEs or serious adverse events (SAEs). Number of participants with treatment-related AEs and SAEs will be reported to sponsor listed in the study report.
Number of participants with abnormal blood routine parameters as assessed by clinical reference values | Day 1 and Day 15
  During the study, blood samples from 2h sample time point will be used for safety check.
  The following parameters will be assessed: AST, ALT, gammaglutamyltransferase, alkaline phosphatase, total cholesterol, low-density lipoprotein- and high-density lipoprotein-cholesterol, triglycerides; creatinine and uric acid. Participants with abnormal values of any of the above-mentioned parameters that fall out of the clinical reference range will be listed and reported.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Menzel, Principal Investigator — BioTeSys GmbH
Locations (1):
- BioTeSys GmbH, Esslingen am Neckar, Germany

IPD SHARING:
Plan to Share IPD: No
Data will not be shared